CLINICAL TRIAL: NCT00188929
Title: Spatio-temporal Response of Non-Hodgkin's Lymphoma to External Beam Radiation Therapy Measuring 18F-Fluorodeoxyglucose (FDG) Uptake Using a Combined PET/CT Scanner: A Pilot Study
Brief Title: Assessment of Treatment Response Using PET/CT Scanner - Non Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Dr. Richard Tsang, Staff Radiation Oncologist, University Health Network, Princess Margaret Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UHN REB 05-0339-C
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2010-08-13 (Estimated); Status verified 2010-08

CONDITIONS: Lymphoma, Non-Hodgkin
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Magnetic Resonance Spectroscopy

INTERVENTIONS:
Procedure: PET Scan with [18F]Fluoro-2-deoxyglucose (FDG)

SUMMARY:
In this study the treatment process will be closely monitored using a novel imaging technology, a PET/CT scanner. PET stands for Positron Emission Tomography and in this case it will be combined with a conventional x-ray Computerized Tomography (CT) scan. This is not a study of any particular form of treatment. The treatment you receive will be the most appropriate standard treatment whether you are in the study or not.

The goal of radiation therapy is to deliver a given amount of radiation dose to the area where there is a lymphoma tumour. We are doing this study to see which part of the tumour reacts to the radiation treatment, and which part does not react, by monitoring the progress of your treatment with a combined PET/CT scan. In particular, changes of the size and shape of the tumour that occur during the treatment can be detected and will be visible on the images. These images will be thoroughly analysed. The ability of the PET/CT scanner to detect these changes during a course of radiation treatment will be the subject of this study. We will also be able to see if this information will eventually relate to or predict whether lymphoma tumours will be completely eradicated by the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of NHL:Any histology
* Stage I-IV
* Measurable disease by CT scan (gross disease measuring at least 2 cm in any one dimension)
* Planned radiation dose prescription >=30 gy, >=20 fractions, >=3weeks duration
* Informed consent
* Previous chemotherapy is allowed, provided the above eligibility criteria are me

Exclusion Criteria:

* To minimize effect from breathing motion, patients presenting with parenchymal lung tumours and tumours involving liver and stomach will be excluded
* Concurrent systemic chemotherapy (glucocorticoids when used alone is allowed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2005-08; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
To quantify spatial and temporal treatment response to radiation therapy in patients with NHL using the co-registered CT and FDG-PET images and assess this response with temporal geometric models.

SECONDARY OUTCOMES:
To assess the feasibility to spatially correlate the abnormalities on the CT image to the FDG uptake on the co-registered PET image using the geometric models.
To determine if the inclusion of a GTV based upon PET images alters (1) the treatment plan based on the initial planning CT; and (2) if GTVs based on CT or PET differ for adaptive plans.
To assess tumor metabolic activity in non-irradiated areas, if detected, and study its temporal changes during a course of radiation treatment (abscopal response).
To link the concentration of the biochemical marker lactate dehydrogenase (LDH) to treatment response.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Tsang, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada